CLINICAL TRIAL: NCT07094672
Title: Development of an Opioid Withdrawal Clinical Outcome Assessment Among Persons With Opioid Use Disorder
Brief Title: Development of an Opioid Withdrawal Clinical Outcome Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kelly Dunn, Director, Kahlert Institute for Addiction Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00114126; UG3DA062907 (NIH)
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder
Keywords: opioid; fentanyl; withdrawal; naloxone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WIthdrawal assessment_precipitated session: Assessment of withdrawal following elicitation
- Withdrawal assessment_spontaneous: Assessment of withdrawal during a period of opioid abstinence

SUMMARY:
Withdrawal management strategies are currently the most utilized and ubiquitous intervention for opioid use disorder in the US, yet existing measures of opioid withdrawal lack Food and Drug Administration (FDA) qualification. This project will develop and validate a clinical outcome assessment (COA) for opioid withdrawal,essential for standardizing withdrawal mitigation strategies and establishing best practices. In line with the FDA's drug development tool qualification guidelines, our methodological process will involve conducting focus groups with persons with lived experience of opioid withdrawal for concept elicitation, refining these concepts through cognitive interviews, and conducting construct and longitudinal validations of the new assessment in laboratory settings and across diverse treatment contexts.

DETAILED DESCRIPTION:
Participants with opioid use disorder will complete a two sessions in a within-subject study design to compare their responses to withdrawal questions after experiencing naloxone-precipitated withdrawal and following an overnight observation of spontaneous withdrawal. All participants will complete both sessions and the order of sessions will be randomized.

The primary outcome will be cognitive interviews, which will be conducted within 8 hours of each observation period ending to query all possible symptoms associated with the withdrawal experience.

Participants will be offered referrals to aftercare prior to study discharge and transitions to treatment programs will be facilitated whenever possible.

ELIGIBILITY:
Inclusion Criteria:

* Past year opioid use disorder, determined by (a) enrollment in current treatment for opioid use disorder and/or (b) an opioid-positive saliva test.
* Fluent in English
* Has experience with opioid withdrawal at least once in the past 30 days

Exclusion Criteria:

* Unable to provide informed consent due to cognitive impairment
* Being pregnant or breastfeeding
* History of psychosis or mania as determined by the MINI
* Exhibiting suicidal behavior in the past 30 days as determined by the C-SSRS
* Circumstances that could interfere with study participation
* Previously participated in affiliated Focus Group study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with opioid use disorder located or able to access the Baltimore regional area
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive interview | Within 8 hours of completing the withdrawal experience
  The experience of withdrawal will be probed qualitatively using cognitive interviews to capture all possible symptoms that opioid withdrawal may elicit in an individual

CONTACTS AND LOCATIONS:
Locations (1):
- Kahlert Institute for Addiction Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data will be qualitative in nature and collapsed into thematic categories. Individualized data will not be shared.